CLINICAL TRIAL: NCT04570969
Title: Improvement of Quality of Life After Live Liver Donation by ESP Peri Operative Analgesia
Brief Title: Benefit of ESP Peri Operative Analgesia for Live Liver Donor Transplantation
Acronym: ESPLIVERDON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vinmec Healthcare System (Other)
Responsible Party: Principal Investigator, Philippe Macaire, Director of anesthesia and pain management - Anesthesiologist MD, Vinmec Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VINMEC LT DON
Record Dates: First submitted 2020-09-20; First posted 2020-09-30 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Liver Transplant Disorder

STUDY DESIGN:
Intervention Model Description: Randomized controlled prospective trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care (No Intervention): Peri-operative analgesia by opioids
- Peri operative regional analgesia (Experimental): Peri-operative analgesia by Continuous bilateral Erector Spinae Catheters
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — Insertion of bilateral catheters in the intersfacia space of erector spinae muscle
  Arms: Peri operative regional analgesia

SUMMARY:
Liver donors have a significant risk to develop persistent and chronic pain around 20 to 30% affecting social and professional life (17%) up to 1 year after the surgery.

To donate a part of liver is a beautiful gift reason why the pain relief must be improved.

Meta-analysis showed that the best prevention against post operative chronic pain are the techniques blocking the pain signal (regional anaesthesia) Patients after liver donation are still in pain even in 2020 with the best multimodal analgesia medications.

Erector sinae Plane Block (ESP) ESP will block the signal and improve the pain relief we hope to demonstrate that it will reduce the risk to develop post operative chronic pain and improve the quality of recovery and the quality of life after liver donation

DETAILED DESCRIPTION:
1. Goals:

   Compare quality of pain relief and quality of life between bilateral ESP bilateral catheters Vs Opioid analgesia in donor patients for liver donation.
2. Methodology:

   • Selection criteria: Age > 18 years old Be volunteer to donate liver Agree to participate in the trial

   • Exclusion criteria: Use of chronic opioids Contra-indication tom perform ESP catheter (Infection near puncture point, Severe thoracic scoliosis, allergie to local anesthestics) A diagnosis of a chronic pain conditionDepression or other psychiatric diagnosis

   • Study design: Prospective Randomized Controlled Trial.

   Patients who agree to join the study will be randomized into 2 groups:

   Group 1 (Control group): standard of care in liver donation : Intraoperative analgesia by Opioid sufentanil and post operative analgesia by PCA opioid morphine Group 2 (treatement group): Standard peri-operative analgesia for liver donation in since Investigators use regional anaesthesia as first line treatement for peri operative analgesia Bilateral ESP catheters with continuous regional analgesia by infusion of local anesthestic (Ropivacaine)

   Sample size: investigators expected to increase the Quality of LIfe (QoL) score (using under-the-curve area) from 36·9 for the ERAS group to 38.3 for ESP group The sample size of 10 patients per group is required to detect such changes assuming a confidence interval of 95% with a power of 90% and alpha = 0.05. Considering 20% of drop-out, the total sample size is 24 patients (12 patients each group)
3. Project outcomes:

   * Primary outcomes Quality of pain relief with opioid consumption
   * Secondary outcomes Duration of hospitalisation participants satisfaction Quality of recovery (QOR 16) Pain at 1 & 3 months rest and mobilization + QOL

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 and less than 61
* Be volunteer to donate liver
* agree to participate to study and consent signed
* Risk of americain society of anesthesiologists score ASA from 1 to 5 score ASA must be 1 only

Exclusion Criteria:

* Use of chronic opioid before the surgery
* A diagnosis of chronic pain condition
* Contra indication to perform ESP catheter
* allergy to local anesthestics
* Depression or psychiatric diagnosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-02-25 (Estimated)

PRIMARY OUTCOMES:
quality of pain relief at rest | from day 0 = day of surgery to day 180
  Visual analgesic score at rest
quality of pain relief at mouvement | from day 0 = day of surgery to day 180
  Visual analgesic score at mouvement

SECONDARY OUTCOMES:
Opioid consumption | from day 0 to 30 days after the day of surgery
  Total dose of opioids required
Duration of hospitalisation | From day = 0 day of the surgery to day to discharge day 15 maximum
  Duration of hospitalisation
Quality of recovery | 1 month after surgery
  Score based on Table quality of recovery including 15 criteria from 0 to 10 each ) = poor 10 = excellent poor recovery scale 0 to 150
Patient satisfaction | 1 month after the surgery
  index from 0 not satisfy to 10 extremely satisfied
Quality of life (QOL) after donation | 1 months and 3 months after surgery
  The Form QOL (36) is a 36-item, patient-reported survey of patient health and mesure the surgical outcomes. The SF-36 is a measure of health status

CONTACTS AND LOCATIONS:
Locations (1):
- VinMec INternational hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No